CLINICAL TRIAL: NCT06628544
Title: The Role of Trained Immunity in Fungal Infection and the Mechanism Behind it
Brief Title: Trained Immunity in Fungal Infection and Its Mechanism
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Zhibing Lu, Professor, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020005
Record Dates: First submitted 2024-09-27; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: BCG Vaccination
Keywords: immunity; metformin; BCG

STUDY DESIGN:
Intervention Model Description: Vaccines (BCG) and Drugs (Metformin)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- BCG vaccination with taking metformin on the day 85 (Experimental)
  Interventions: Biological: BCG vaccination; Drug: Metformin is administered on the day 85
- BCG vaccination without metformin (Experimental)
  Interventions: Biological: BCG vaccination
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- BCG vaccination with taking metformin on the day 0 (Experimental)
  Interventions: Biological: BCG vaccination; Drug: Metformin is administered on the day 0
- BCG vaccination with taking metformin on the day 9 (Experimental)
  Interventions: Biological: BCG vaccination; Drug: Metformin is administered on the day 9

INTERVENTIONS:
Biological: BCG vaccination — BCG vaccination
  Arms: BCG vaccination with taking metformin on the day 0; BCG vaccination with taking metformin on the day 85; BCG vaccination with taking metformin on the day 9; BCG vaccination without metformin
Drug: Metformin is administered on the day 0 — Metformin is administered on the day 0
  Arms: BCG vaccination with taking metformin on the day 0
Other: Placebo — Placebo
  Arms: Placebo
Drug: Metformin is administered on the day 9 — Metformin is administered on the day 9
  Arms: BCG vaccination with taking metformin on the day 9
Drug: Metformin is administered on the day 85 — Metformin is administered on the day 85
  Arms: BCG vaccination with taking metformin on the day 85

SUMMARY:
Investigator vaccinated 76 healthy BCG-naive participant with BCG, while 3 participants received. Half of BCG-vaccinated participants (n = 38) received an incremental dose of metformin for 6 days (up to 1,000 mg twice daily on day 6). On the day 0 (total 20; n = 10 for BCG vaccination, n = 10 for BCG vaccination plus taking metformin), day 14 (total 30; n=15 for BCG vaccination, n = 15 for BCG vaccination plus taking metformin), day 90 (total 26; n = 13 for BCG vaccination, n=13 for BCG vaccination plus taking metformin) of BCG vaccination, PBMCs were isolated, restimulated with C. albicans or Mycobacterium tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy BCG-naive participants.
* The ages range from 20 to 45.
* Participants without any infections or immune deficiencies.

Exclusion Criteria:

* Participants when infections or other illnesses occurred during the clinical trial.
* Participants who have a fever of unknown causes during the clinical trial.
* Participants who have gotten other vaccines during the clinical trial.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The level of IL-6 | Five days of continuous medication+24 hours restimulation of C.albicans or Mycobacterium tuberculosis
  After 5 days of continuous medication, PBMCs were isolated, restimulated with C. albicans or Mycobacterium tuberculosis. And the level of cytokines were determined by Elisa.
The level of TGF-alpha | Five days of continuous medication+24 hours restimulation of C.albicans or Mycobacterium tuberculosis
  After 5 days of continuous medication, PBMCs were isolated, restimulated with C. albicans or Mycobacterium tuberculosis. And the level of cytokines were determined by Elisa.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan University, Wuhan, Hubei, China, China

IPD SHARING:
Plan to Share IPD: No